CLINICAL TRIAL: NCT01031225
Title: A Non-Randomized, Open-label, Multi-Center, Multi-Cohort Phase 2 Study Evaluating the Efficacy and Safety of STA-9090 in Subjects With Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: A Study of the HSP90 Inhibitor, STA-9090 in Subjects With Stage IIIB or IV Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9090-06
Record Dates: First submitted 2009-11-16; First posted 2009-12-14 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Synta; STA 9090; ganetespib); Lung Cancer; Non Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: STA 9090

INTERVENTIONS:
Drug: STA 9090 — STA-9090 IV infusion once per week for three consecutive weeks followed by a 1 week dose-free interval

SUMMARY:
This is a phase 2 study of the HSP90 inhibitor, STA-9090 (ganetespib) in subjects with stage IIIB or IV non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of Stage IIIB (with pleural effusion) or Stage IV NSCLC with measurable disease by RECIST and evidence of progression
* Availability of tissue for analysis
* ECOG Performance Status 0 or 1
* Adequate organ function as defined in the protocol.
* Must be at least 18 years old and able and willing to sign a written informed consent document

Exclusion Criteria:

* Poor venous access requiring an indwelling catheter for study drug administration
* Women who are pregnant or lactating
* Ventricular ejection fraction < or = to 55% at baseline
* Any uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-11; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival rate | 16 weeks

SECONDARY OUTCOMES:
Objective Response Rate, Disease Control Rate, Progression Free Survival, Overall Survival | 18 months
Safety and tolerability as measured by adverse event rates and laboratory evaluations | 16 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Arizona Cancer Center; University of Arizona, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - City of Hope Medical Center, Duarte, California
  - UCLA Health System, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Emory University- Winship Cancer Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of North Carolina, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington